CLINICAL TRIAL: NCT03380130
Title: A Multicenter, Open-label, Single-arm Study of the Safety and Antitumoral Efficacy of Nivolumab After SIRT Using SIR-Spheres for the Treatment of Patients With HepatoCellular Carcinoma That Are Candidates for Locoregional Therapies
Brief Title: A Study of the Safety and Antitumoral Efficacy of Nivolumab After SIRT for the Treatment of Patients With HCC
Acronym: NASIR-HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Sirtex Medical (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NASIR-HCC/CA209-992
Record Dates: First submitted 2017-10-20; First posted 2017-12-20 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Liver cancer; Hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIRT and Nivolumab (Experimental): SIRT (selective internal radiation therapy) will be performed in a single session using SIR-Spheres resin microspheres. After 3 weeks, nivolumab 240 mg every 2 weeks will be initiated
  Interventions: Drug: Nivolumab; Device: SIR-Spheres

INTERVENTIONS:
Drug: Nivolumab — An anti-programmed death 1 monoclonal antibody
  Other Names: Opdivo
Device: SIR-Spheres — Resin microspheres labeled with the radioactive isotope yttrium 90 that serves as a source of beta radiation
  Other Names: radioembolization, transarterial radioembolization (TARE)

SUMMARY:
The purpose of this study is to evaluate the effect of the anti-programmed death 1 (PD-1) agent nivolumab following selective internal radiation therapy (SIRT) for patients with unresectable hepatocellular carcinoma (HCC).

SIRT using yttrium90-loaded microspheres is increasingly used to treat patients with HCC, particularly those that are not good candidates for transarterial chemoembolization or TACE. SIRT induces disease control (objective tumor remission or stabilization) in most patients while progression usually results from the growth of new lesions. SIR-Spheres are resin-made microspheres used for SIRT.

On the other hand, nivolumab is under clinical development for the treatment of more advanced HCC. Available data in patients that mostly had progression to other therapies and vascular involvement or metastatic disease show significant systemic antitumor activity that results in durable objective remissions and disease stabilizations.

Therefore, in patients with HCC that has not spread beyond the liver, the systemic action of nivolumab may improve the anti-tumor effect of SIRT. Furthermore, by inducing immunogenic tumor cell death, SIRT may have a synergistic effect with nivolumab.

DETAILED DESCRIPTION:
Worldwide, intra-arterial therapies are the mainstay of the treatment of patients with HCC in the intermediate stage or in the advanced stage because of portal vein invasion. While transarterial chemoembolization (TACE) is the most widely applied intra-arterial therapy, not all patients in the intermediate stage are good candidates for this procedure and TACE is formally contraindicated in the presence of portal vein invasion. Selective Internal Radiation Therapy (SIRT) using yttrium90-loaded microspheres is increasingly used to treat such patients that are not good candidates for TACE. SIR-Spheres are resin-made microspheres extensively used for SIRT and there is consistent level 2 evidence of its activity in HCC. SIRT induces disease control (partial objective remission or tumor stabilization) in the majority of patients while progression usually results from the growth of new lesions.

Nivolumab is under clinical development for the treatment of advanced stage HCC. Preliminary data in a population that mostly had progression to other therapies, vascular involvement or metastatic disease suggest significant systemic antitumor activity that results in durable objective remissions and disease stabilizations. In patients with HCC that has not spread beyond the liver, the systemic action of nivolumab may improve the anti-tumor effect of SIRT by providing eradication or sustained tumor growth control of residual disease in treated lesions and other locations (intrahepatic or extrahepatic micrometastasis). Furthermore, by inducing immunogenic tumor cell death, SIRT may have a synergistic effect with immune checkpoint inhibitors including nivolumab. Besides, SIRT and nivolumab are by and large well tolerated. The sequential use of SIRT and nivolumab could have strong antitumor activity and a favorable safety profile and therefore deserves to be tested in patients with intermediate to advanced tumor stages.

The primary objective of the study is therefore to evaluate the safety of nivolumab in combination with SIRT using SIR-Spheres. The secondary objective is to evaluate the anti-tumor activity of nivolumab in combination with SIRT using SIR-Spheres. Exploratory objectives are to evaluate the role of blood and tissue biomarkers in determining the anti-tumor activity of nivolumab in combination with SIRT using SIR-Spheres; to evaluate the utility of baseline or on-treatment soluble markers that may serve as surrogate markers of efficacy; and to explore the role of the ALBI score in predicting patient outcomes.

SIRT will be performed as a single-day treatment using SIR-Spheres resin microspheres as detailed in Gil-Alzugaray et al. 2013. Three weeks after SIRT, patients will start receiving nivolumab every 2 weeks until completion of 8 courses of 3 bi-weekly nivolumab doses, toxicity, or tumor progression defined using RECIST 1.1 criteria. Patients will be allowed to continue nivolumab treatment beyond progression under strict protocol-defined circumstances. All subjects will undergo tumor assessments at every q6 week for the first year, and then q12 week thereafter until radiographic progression. Patients will complete a follow-up Visit 100 days from the last dose of nivolumab and will then be followed for overall survival.

Patients with all etiologies could be recruited. Those with chronic hepatitis B will be on antiviral therapy per regional standard of care guidelines. Patients with chronic hepatitis C may receive treatment for this condition with direct antiviral agents during the treatment period as per local practice guidelines.

A tumor sample obtained before SIRT and blood samples obtained before SIRT and before and after nivolumab will be used for correlative biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC based on histology or non-invasive criteria if cirrhotics. Patients with fibrolamellar carcinoma are not excluded.
* Cirrhosis absent, non-viral or due to hepatitis C or B virus infection. Subjects with chronic hepatitis B virus infection must be on effective antiviral therapy
* Preserved liver function (without cirrhosis or with compensated cirrhosis in Child Pugh Class A).
* ECOG performance status 0 or 1
* Willing to have a liver biopsy pre-treatment
* Considered candidates for locoregional therapy using SIR-Spheres based on

  * the absence of extrahepatic disease (patients with regional lymph nodes < 2 cm in short axis are accepted)
  * unsuitability for liver resection or transplantation, or percutaneous ablation
  * considered not good candidates for TACE because they have; Single tumors larger than 5 cm. Multiple tumors that cannot be targeted superselectively. Unilobar tumors with segmental or lobar portal vein thrombosis.
* At least one measurable lesion by RECIST 1.1 criteria.
* Adequate organ and marrow function as evidenced by:

  * White blood cell count ≥ 2000/μL.
  * Neutrophils ≥ 1000/μL.
  * Platelets ≥ 60 x 103/μL.
  * Hemoglobin ≥ 9.0 g/dL.
  * Creatinine Clearance > 40 mL/min.
  * AST and ALT ≤ 5 X ULN
  * Bilirubin ≤ 2 mg/dL
  * INR ≤ 1.8.
  * Albumin ≥ 3.0 g/dL
* Willing and able to comply with immune-monitoring sample collection and required study follow-up.

Exclusion Criteria:

* Any history of hepatic encephalopathy
* Any prior (within 6 months) or current clinical ascites.
* Any history of clinically meaningful variceal bleeding within the last three months.
* Active coinfection with both hepatitis B and C or hepatitis D infection in subjects with hepatitis B
* Occlusive main trunk portal vein thrombosis or absence of intrahepatic portal blood flow if patient carries a portocaval shunt.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
* Any autoimmune disease that may require immunosuppressive therapy.
* Any severe organ disease
* Prior therapy with any drug specifically targeting T-cell costimulation or checkpoint pathways.
* Prior organ allograft or allogeneic bone marrow transplantation
* Active bacterial or fungal infections within 7 days of study entry.
* Any condition requiring systemic treatment with corticosteroids or other immunosuppressive medications within 14 days of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Rate and type of adverse events, liver decompensation, and transient and permanent drug discontinuations due to toxicity. | Two years
  The incidence of observed adverse events (AE) will be evaluated according to NCI CTCAE version 4.03. Particular attention will be given to adverse events that may follow enhanced T cell activation (hepatitis, dermatitis, colitis, pneumonitis, endocrinopathy or other immune-mediated AEs) and radiation damage to non-target organs (REILD, radiation pneumonitis and GI ulcers).

SECONDARY OUTCOMES:
Response rate | Two years
Disease control rate | Two years
Duration of response | From date of complete or partial response to the date of progression, assessed up to 36 months.
Time to progression | From date of SIRT to the date of progression, assessed up to 36 months.
Progression-free survival | From date of SIRT to the date of progression or death, whichever came first, assessed up to 36 months.
Overall survival | From date of SIRT to the date of death, assessed up to 36 months
Pattern of progression according to RECIST 1.1 criteria. | Two years
  Event that trigers the evaluation of tumor assessment as progressive disease according to RECIST 1.1 criteria, subclassified as 1) growth of existing tumor lesions only; 2) occurrence of new lesions inside the liver irrespective of previous criterion; and 3) occurrence of new lesions outside the liver irrespective of the two prior criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Sangro, MD, Principal Investigator — Liver Unit, Clínica Universidad de Navarra
Locations (9):
- Spain (9):
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Clinic, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangro B, Salem R. Transarterial chemoembolization and radioembolization. Semin Liver Dis. 2014 Nov;34(4):435-43. doi: 10.1055/s-0034-1394142. Epub 2014 Nov 4. PMID 25369305
- [Background] Bolondi L, Burroughs A, Dufour JF, Galle PR, Mazzaferro V, Piscaglia F, Raoul JL, Sangro B. Heterogeneity of patients with intermediate (BCLC B) Hepatocellular Carcinoma: proposal for a subclassification to facilitate treatment decisions. Semin Liver Dis. 2012 Nov;32(4):348-59. doi: 10.1055/s-0032-1329906. Epub 2013 Feb 8. PMID 23397536
- [Background] Sangro B, Carpanese L, Cianni R, Golfieri R, Gasparini D, Ezziddin S, Paprottka PM, Fiore F, Van Buskirk M, Bilbao JI, Ettorre GM, Salvatori R, Giampalma E, Geatti O, Wilhelm K, Hoffmann RT, Izzo F, Inarrairaegui M, Maini CL, Urigo C, Cappelli A, Vit A, Ahmadzadehfar H, Jakobs TF, Lastoria S; European Network on Radioembolization with Yttrium-90 Resin Microspheres (ENRY). Survival after yttrium-90 resin microsphere radioembolization of hepatocellular carcinoma across Barcelona clinic liver cancer stages: a European evaluation. Hepatology. 2011 Sep 2;54(3):868-78. doi: 10.1002/hep.24451. Epub 2011 Jun 30. PMID 21618574
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Gil-Alzugaray B, Chopitea A, Inarrairaegui M, Bilbao JI, Rodriguez-Fraile M, Rodriguez J, Benito A, Dominguez I, D'Avola D, Herrero JI, Quiroga J, Prieto J, Sangro B. Prognostic factors and prevention of radioembolization-induced liver disease. Hepatology. 2013 Mar;57(3):1078-87. doi: 10.1002/hep.26191. Epub 2013 Feb 15. PMID 23225191
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Derived] De la Torre-Alaez M, Matilla A, Varela M, Inarrairaegui M, Reig M, Lledo JL, Arenas JI, Lorente S, Testillano M, Marquez L, Iserte G, Argemi J, Gomez-Martin C, Rodriguez-Fraile M, Bilbao JI, Pollock RF, Pohlmann J, Agirrezabal I, Sangro B. Health-related quality of life in patients with unresectable hepatocellular carcinoma treated with SIRT and nivolumab: a sub-analysis of the NASIR-HCC trial. J Patient Rep Outcomes. 2025 Apr 8;9(1):39. doi: 10.1186/s41687-025-00873-6. PMID 40198533
- [Derived] de la Torre-Alaez M, Matilla A, Varela M, Inarrairaegui M, Reig M, Lledo JL, Arenas JI, Lorente S, Testillano M, Marquez L, Da Fonseca L, Argemi J, Gomez-Martin C, Rodriguez-Fraile M, Bilbao JI, Sangro B. Nivolumab after selective internal radiation therapy for the treatment of hepatocellular carcinoma: a phase 2, single-arm study. J Immunother Cancer. 2022 Nov;10(11):e005457. doi: 10.1136/jitc-2022-005457. PMID 36450386
- [Derived] Ezponda A, Rodriguez-Fraile M, Morales M, Vivas I, De La Torre M, Sangro B, Bilbao JI. Hepatic Flow Redistribution is Feasible in Patients with Hepatic Malignancies Undergoing Same-Day Work-Up Angiography and Yttrium-90 Microsphere Radioembolization. Cardiovasc Intervent Radiol. 2020 Jul;43(7):987-995. doi: 10.1007/s00270-019-02371-x. Epub 2019 Dec 17. PMID 31848672